CLINICAL TRIAL: NCT02782468
Title: A Phase 1/1b, Open-label Study of Pevonedistat (MLN4924, TAK-924) as Single Agent and in Combination With Azacitidine in Adult East Asian Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Pevonedistat in Adult East Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pevonedistat-1012; U1111-1166-8630 (Other: WHO)
Record Dates: First submitted 2016-05-20; First posted 2016-05-25 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-01

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: Drug Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — pevonedistat; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1, Cohort 1: Pevonedistat 25 mg/m^2 (Experimental): Pevonedistat, 25 milligram per square meter (mg/m^2), 60-minute infusion, intravenously, on Days 1, 3 and 5, followed by a rest period of 16 days, in 21-day treatment cycles.
  Interventions: Drug: Pevonedistat 25 mg/m^2
- Arm 1, Cohort 2: Pevonedistat 44 mg/m^2 (Experimental): Pevonedistat, 44 mg/m^2, 60-minute infusion, intravenously, on Days 1, 3, and 5, followed by a rest period of 16 days, in 21-day treatment cycles.
  Interventions: Drug: Pevonedistat 44 mg/m^2
- Arm 2, Cohort 1: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 (Experimental): Pevonedistat 10 mg/m^2, 60-minute infusion, intravenously, on Days 1, 3, and 5 and azacitidine 75 mg/m^2, on Days 1 to 5, and Days 8 and 9, intravenously or subcutaneously, followed by a rest period of 19 days, in 28-day treatment cycles.
  Interventions: Drug: Pevonedistat 10 mg/m^2; Drug: Azacitidine 75 mg/m^2
- Arm 2, Cohort 2: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2 (Experimental): Pevonedistat 20 mg/m^2, 60-minute infusion, intravenously, on Days 1, 3, and 5 and azacitidine 75 mg/m^2, on Days 1 to 5, and Days 8 and 9, intravenously or subcutaneously, followed by a rest period of 19 days, in 28-day treatment cycles.
  Interventions: Drug: Pevonedistat 20 mg/m^2; Drug: Azacitidine 75 mg/m^2

INTERVENTIONS:
Drug: Pevonedistat 25 mg/m^2 — Pevonedistat 25 mg/m^2 intravenous infusion.
  Arms: Arm 1, Cohort 1: Pevonedistat 25 mg/m^2
Drug: Pevonedistat 44 mg/m^2 — Pevonedistat 44 mg/m^2 intravenous infusion.
  Arms: Arm 1, Cohort 2: Pevonedistat 44 mg/m^2
Drug: Pevonedistat 10 mg/m^2 — Pevonedistat 10 mg/m^2 intravenous infusion.
  Arms: Arm 2, Cohort 1: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2
Drug: Pevonedistat 20 mg/m^2 — Pevonedistat 20 mg/m^2 intravenous infusion.
  Arms: Arm 2, Cohort 2: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Drug: Azacitidine 75 mg/m^2 — Azacitidine 75 mg/m^2 intravenous or subcutaneous formulation.
  Arms: Arm 2, Cohort 1: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2; Arm 2, Cohort 2: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of pevonedistat administered as a single agent and in combination with azacitidine in adult east Asian participants with acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
The drug being tested in this study is called Pevonedistat. Pevonedistat is being tested to treat people with myelodysplastic syndromes MDS (including nonproliferative chronic myelomonocytic leukemia [CMML]) and AML (acute myeloid leukaemia) as a single-agent and in combination treatment with azacitidine. This study will look at the safety and tolerability, the recommended phase 2/phase 3 dose of pevonedistat administered in combination with azacitidine, pharmacokinetics and response to treatment in participants who take single agent pevonedistat compared to participants who take pevonedistat and azacitidine.

The study will enroll approximately 37 participants. Participants will be assigned into one of the four treatment groups which will remain disclosed to the patient and study doctor during the study. Participants will be first enrolled at single-agent low dose level (25 mg/m^2). If this dose is tolerable, participants will be enrolled in parallel at single-agent higher dose level (44 mg/m^2) and in combination treatment cohorts.

* Pevonedistat 25 mg/m^2
* Pevonedistat 44 mg/m^2
* Pevonedistat 10 mg/m^2 and azacitidine 75 mg/m^2 combination
* Pevonedistat 20 mg/m^2 and azacitidine 75 mg/m^2 combination Participants will receive pevonedistat infusion intravenously and azacitidine via intravenous or subcutaneous route.

This multi-center trial will be conducted in Japan, Korea and Taiwan. The overall time to participate in this study is approximately 24 months. Participants will attend the End of Study (EOS) visit for safety, 30 days after receiving their last dose of study drug or before the start of subsequent antineoplastic therapy (other than hydroxyurea).

ELIGIBILITY:
Inclusion Criteria include, in part:

1. East Asian patients aged 18 years or older (or minimum age of legal consent consistent with local regulations) when written study informed consent is obtained must meet 1 of the following diagnosis criteria for either the Single-Agent Arm or the Combination Arm (additional restrictions apply to the Single Agent Arm):

   a. Are male and female participants with WHO-defined AML, including leukemia secondary to prior chemotherapy or resulting from an antecedent hematologic disorder, who have failed to achieve CR or who have relapsed after prior therapy (R/R) and are not candidates for potentially curative treatment, or ii. Are male and female participants aged 60 years or older with previously untreated AML who have bone marrow blasts <30% and who are not candidates for standard induction chemotherapy, or iii. Are male and female participants with WHO-defined MDS that meets the IPSS-R criteria for the very high, high, or intermediate risk group, for whom standard curative, life-prolonging treatment does not exist or is no longer effective (R/R), or iv. Are male and female participants with previously untreated MDS that meets the IPSS-R criteria for the very high, high, or intermediate risk group, or vi. Are male and female participants with WHO-defined CMML-2 or CMML-1 that meets the IPSS-R criteria for the very high, high, or intermediate risk group CMML-1 participants must have bone marrow blasts >=5%
2. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Able to undergo bone marrow aspiration and biopsy at Screening.

Exclusion Criteria include, in part:

1. Acute promyelocytic leukemia (as diagnosed by morphologic examination of bone marrow, by fluorescent in situ hybridization or cytogenetics [t (15:17)] of peripheral blood or bone marrow, or by other accepted analysis) or AML associated with t (9;22) karyotypes or molecular.
2. More than 3 prior lines of therapy (Combination Arm only).
3. Prior therapy with hypomethylating agents (example, azacitidine, decitabine). (Combination Arm only).
4. Is eligible for a hematopoietic stem cell transplant.
5. Is a female participant who is lactating and breastfeeding or who have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
6. Had treatment with any investigational products within 14 days before the first dose of any study drug.
7. Has known hypersensitivity to azacitidine or mannitol (Combination Arm only).
8. Has known central nervous system involvement.
9. Had systemic antineoplastic therapy or radiotherapy within 14 days before the first dose of any study drug, except for hydroxyurea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- Japan (4):
  - Maebashi
  - Nagoya
  - Sendai
  - Tokyo
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Jeonnam
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Handa H, Cheong JW, Onishi Y, Iida H, Kobayashi Y, Kim HJ, Chiou TJ, Izutsu K, Tsukurov O, Zhou X, Faessel H, Yuan Y, Sedarati F, Faller DV, Kimura A, Wu SJ. Pevonedistat in East Asian patients with acute myeloid leukemia or myelodysplastic syndromes: a phase 1/1b study to evaluate safety, pharmacokinetics and activity as a single agent and in combination with azacitidine. J Hematol Oncol. 2022 May 11;15(1):56. doi: 10.1186/s13045-022-01264-w. PMID 35545778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Japan, Taiwan and South Korea from 16 May 2016 to 25 January 2022.
Pre-assignment Details: Participants with a historical diagnosis of relapsed/refractory (R/R) acute myeloid leukemia (AML) or R/R higher risk (HR) myelodysplastic syndromes (MDS) (including nonproliferative chronic myelomonocytic leukemia [CMML]) were enrolled to receive single agent pevonedistat or combination of pevonedistat and azacitidine.
Groups:
- Single Agent Arm: Pevonedistat 25 mg/m^2: Pevonedistat 25 milligram per square meter (mg/m^2), infusion, intravenously, on Days 1, 3 and 5, followed by a rest period of 16 days, in each 21-day treatment cycle until disease progression or symptomatic deterioration.
- Single Agent Arm: Pevonedistat 44 mg/m^2: Pevonedistat 44 mg/m^2, infusion, intravenously, on Days 1, 3, and 5, followed by a rest period of 16 days, in each 21-day treatment cycle until disease progression or symptomatic deterioration.
- Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2: Pevonedistat 10 mg/m^2, infusion, intravenously, on Days 1, 3, and 5 along with azacitidine 75 mg/m^2, injection, intravenously in Cycle 1 and intravenously or subcutaneously from Cycle 2 onwards, on Days 1 to 5, and Days 8 and 9, followed by a rest period of 19 days, in each 28-day treatment cycle until disease progression or symptomatic deterioration.
- Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2: Pevonedistat 20 mg/m^2, infusion, intravenously, on Days 1, 3, and 5 along with azacitidine 75 mg/m^2, injection, intravenously in Cycle 1 and intravenously or subcutaneously from Cycle 2 onwards, on Days 1 to 5, and Days 8 and 9, followed by a rest period of 19 days, in each 28-day treatment cycle until disease progression or symptomatic deterioration.
Period: Overall Study
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Started | 3 | 7 | 3 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 3 | 10
Not completed — Progressive Disease | 2 | 5 | 0 | 4
Not completed — Adverse Event | 0 | 2 | 2 | 3
Not completed — Other | 0 | 0 | 1 | 1
Not completed — Initiation of Hematopoietic Stem Cell Transplant | 0 | 0 | 0 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all enrolled participants who received at least 1 dose of any study drug, pevonedistat or azacitidine.
Groups:
- Single Agent Arm: Pevonedistat 25 mg/m^2: Pevonedistat 25 mg/m^2, infusion, intravenously, on Days 1, 3 and 5, followed by a rest period of 16 days, in each 21-day treatment cycle until disease progression or symptomatic deterioration.
- Total: Total of all reporting groups
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 3 | 7 | 3 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (5.20) | 69.0 (11.27) | 65.0 (9.54) | 64.9 (8.52) | 67.9 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 3 | 4
  Male | 2 | 7 | 3 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 3 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 3 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 2 | 2 | 1 | 7 | 12
  Korea, South | 1 | 2 | 0 | 1 | 4
  Taiwan | 0 | 3 | 2 | 2 | 7
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] | 1.5 (0.26) | 1.7 (0.21) | 1.7 (0.04) | 1.7 (0.18) | 1.7 (0.20)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose through 30 days after the last dose of study drug: single agent arms (up to Cycle 19 [up to Day 429]) (Cycle=21 days); combination arms (up to Cycle 65 [up to Day 1850]) (Cycle=28 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 10
Participants
  TEAEs | 3 | 7 | 3 | 10
  SAEs | 2 | 7 | 3 | 6

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 During Cycle 1
Description: DLT: Any of following events considered possibly related to study drug(s) by investigator: Grade (G) 3 or greater nausea and/or emesis despite use of optimal antiemetic prophylaxis; G3 diarrhea occurred despite maximal supportive therapy; G3 arthralgia/myalgia despite use of optimal analgesia; G3 nonhematologic toxicity with exceptions: 1) Brief fatigue, 2) hypophosphatemia; Persistent elevations of transaminases/bilirubin above G2 beyond 2 days between doses; Other study drug-related nonhematologic toxicities G2 or greater, required a dose reduction/discontinuation of pevonedistat. G3 or greater hematologic toxicities, including G3 or 4 febrile neutropenia, considered DLTs if: A delay in initiation of Cycle 2 due to lack of adequate recovery from treatment-related toxicity: 1) Of more than (>) 4 weeks due to hematologic toxicity believed not related to leukemic infiltration. Bone marrow (BM) evaluation may have been required. 2) Of >2 weeks due to nonhematologic toxicities.
Time Frame: Cycle 1 (Cycle length = 21 days [single agent arms]; 28 days [combination arms])
Population: The DLT evaluable population was defined as all participants who either experienced DLT during Cycle 1 or received all scheduled doses of study drug during Cycle 1 without DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 6 | 3 | 8
Participants | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Time Frame: Baseline up to Cycle 19 (up to Day 399) in single agent arms (Cycle=21days) and Cycle 65 (up to Day 1820) in combination arms (Cycle=28 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 10
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Pevonedistat When Administered Alone and in Combination With Azacitidine on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1: pre-infusion and at multiple time points (up to 48 hours) post-infusion (Cycle length = 21 days [single agent arms]; 28 days [combination arms])
Population: Pharmacokinetic (PK) evaluable population was defined as all enrolled participants who had sufficient dosing in Cycle 1 and pevonedistat concentration-time data to reliably estimate PK parameters by noncompartmental analysis methods and who had not received any excluded concomitant medications per the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 10
nanogram per milliliter (ng/mL) | 253 (37.6) | 410 (45.5) | 67.0 (5.9) | 160 (25.7)

5. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Pevonedistat When Administered Alone and in Combination With Azacitidine on Cycle 1 Day 5
Time Frame: Cycle 1 Day 5: pre-infusion and at multiple time points (up to 48 hours) post-infusion (Cycle length = 21 days [single agent arms]; 28 days [combination arms])
Population: PK evaluable population was defined as all enrolled participants who had sufficient dosing in Cycle 1 and pevonedistat concentration-time data to reliably estimate PK parameters by noncompartmental analysis methods and who had not received any excluded concomitant medications per the protocol. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 8
ng/mL | 252 (9.9) | 453 (38.7) | 76.1 (17.6) | 170 (33.7)

6. Primary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Pevonedistat When Administered Alone and in Combination With Azacitidine on Cycle 1 Day 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 8
hour*nanogram per milliliter (h*ng/mL) | 1515 (9.1) | 2163 (25.7) | 647 (41.3) | 1224 (14.9)

7. Primary Outcome: CL: Total Clearance for Pevonedistat When Administered Alone and in Combination With Azacitidine on Cycle 1 Day 1
Time Frame: as for outcome 4
Population: PK evaluable population was defined as all enrolled participants who had sufficient dosing in Cycle 1 and pevonedistat concentration-time data to reliably estimate PK parameters by noncompartmental analysis methods and who had not received any excluded concomitant medications per the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 10
liter per hour | 24.1 (20.1) | 32.6 (41.7) | 22.8 (48.8) | 28.4 (23.9)

8. Primary Outcome: CL: Total Clearance for Pevonedistat When Administered Alone and in Combination With Azacitidine on Cycle 1 Day 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 7 | 3 | 8
liter per hour | 24.0 (23.0) | 34.8 (34.6) | 28.1 (38.3) | 28.9 (23.7)

9. Secondary Outcome: Overall Response Rate (ORR) for Participants With AML
Description: ORR for AML was defined as the percentage of participants with a complete remission (CR), CR with incomplete blood count recovery (CRi), or partial remission (PR) based on Modified International Working Group (IWG) Response Criteria for AML. CR was defined as participant achieved the morphologic leukemia-free state and had an absolute neutrophil count (ANC) of more than 1,000 per microliter (/mcL) and platelets of greater than or equal to (>=) 100,000/mcL. A morphologic leukemia-free state requires less than (<) 5 percent (%) blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. CRi was, after chemotherapy, some participants who fulfilled all of the criteria for CR except for residual neutropenia (<1,000/mcL) or thrombocytopenia (<100,000/mcL). PR designation required all the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to between 5% and 25% in the bone marrow aspirate.
Time Frame: From first dose up to 30 days after last dose of study drug or before start of subsequent antineoplastic therapy, whichever comes earlier up to Cycle 19 (up to Day 429, single agent)(Cycle=21 days) and Cycle 65 (up to Day 1850, combination)(Cycle=28 days)
Population: Response evaluable population was defined as all participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 post baseline disease assessment. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 2 | 5
percentage of participants | 0 | 0 | 50 | 80

10. Secondary Outcome: ORR for Participants With MDS
Description: ORR for MDS: Percentage of participants with CR,PR or hematologic improvement(HI) based on IWG Response Criteria. CR: BM:<=5% myeloblasts with normal maturation of all cell lines; persistent dysplasia noted peripheral blood: hemoglobin (Hgb)>=11 gram per deciliter (g/dL),platelets>=100*10^9/L,neutrophils >=1.0*10^9/L, blasts 0%. PR:CR criteria if abnormal before treatment except: BM blasts decreased by >=50% from pretreatment but still>5%; cellularity, morphology not relevant. HI criteria: Erythroid response:Hgb up by >=1.5 g/dL; transfused RBC reduced by at least 4 red blood cell (RBC) transfusions/8 weeks comparatively last 8 weeks; Platelet response: Increase of >=30*10^9/L for participants starting with >20*10^9/L platelets; increase from <20*10^9/L to >20*10^9/L and by 100%; Neutrophil response: At least 100% and absolute increase >0.5*10^9/L; Progression/relapse after HI: Granulocytes/platelets decreased by 50% from maximum; Hgb reduced by >=1.5 g/dL; transfusion dependence.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 0 | 2 | 1 | 3
percentage of participants |  | 0 | 100 | 0

11. Secondary Outcome: Percentage of Participants With CR for Participants With AML
Description: CR was defined as participant achieved the morphologic leukemia-free state and had an ANC of more than 1,000/mcL and platelets of >=100,000/mcL. A morphologic leukemia-free state requires <5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. CR assessment was based on IWG Response Criteria.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 2 | 5
percentage of participants | 0 | 0 | 50 | 0

12. Secondary Outcome: Percentage of Participants With CR for Participants With MDS
Description: CR was defined as participant with bone marrow: less than or equal to (<=) 5% myeloblasts with normal maturation of all cell lines; persistent dysplasia was noted peripheral blood: Hgb >=11 g/dL, platelets >=100*10^9/L, neutrophils >=1.0*10^9 per liter (/L), blasts 0%. CR assessment was based on IWG Response Criteria.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2+ Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2+ Azacitidine 75 mg/m^2
Number analyzed (Participants) | 0 | 2 | 1 | 3
percentage of participants |  | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started after first dose through 30 days after the last dose of study drug: single agent arms (up to Cycle 19 [up to Day 429]) (Cycle=21 days); combination arms (up to Cycle 65 [up to Day 1850]) (Cycle=28 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Combination Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2: Pevonedistat 10 mg/m^2, infusion, intravenously, on Days 1, 3, and 5 along with azacitidine 75 mg/m^2, injection, intravenously in Cycle 1 and intravenously or subcutaneously from Cycle 2 onwards, on Days 1 to 5, and Days 8 and 9, followed by a rest period of 19 days, in each 28-day treatment cycle until disease progression or symptomatic deterioration.
- Combination Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2: Pevonedistat 20 mg/m^2, infusion, intravenously, on Days 1, 3, and 5 along with azacitidine 75 mg/m^2, injection, intravenously in Cycle 1 and intravenously or subcutaneously from Cycle 2 onwards, on Days 1 to 5, and Days 8 and 9, followed by a rest period of 19 days, in each 28-day treatment cycle until disease progression or symptomatic deterioration.
Arm/Group | Single Agent Arm: Pevonedistat 25 mg/m^2 | Single Agent Arm: Pevonedistat 44 mg/m^2 | Combination Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Combination Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/7 | 1/3 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 7/7 | 3/3 | 6/10
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Arm: Pevonedistat 25 mg/m^2 (N=3) | Single Agent Arm: Pevonedistat 44 mg/m^2 (N=7) | Combination Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 (N=3) | Combination Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 (N=10)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 5 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Arm: Pevonedistat 25 mg/m^2 (N=3) | Single Agent Arm: Pevonedistat 44 mg/m^2 (N=7) | Combination Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 (N=3) | Combination Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 (N=10)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 3
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Arterial fibrosis (Vascular disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 3
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Bacillus bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 4
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1
Catheter site extravasation (General disorders) | 0 | 0 | 0 | 1
Catheter site injury (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 1
Catheter site swelling (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival pallor (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 2 | 7
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 3
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Enlarged uvula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 3
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2
Hypotension (Vascular disorders) | 0 | 2 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 1 | 2
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 2 | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 3
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Penis injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 1 | 2
Platelet count decreased (Investigations) | 0 | 1 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pustule (Infections and infestations) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 4 | 1 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 3
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 6
Weight decreased (Investigations) | 0 | 2 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT02782468/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02782468/SAP_001.pdf